CLINICAL TRIAL: NCT03334981
Title: Interest of Concentrations in Meconium of Drugs Used for Treatment of Pregnant Opioid-dependent Woman as a Prognostic Factor of Time, Severity and Duration of Neonatal Abstinence Syndrome
Brief Title: Interest of Concentrations in Meconium of Buprenorphine and Methadone as a Prognostic Factor of NAS Outcome
Acronym: SUBOPGEST
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 11-061
Record Dates: First submitted 2016-09-07; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2016-10

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: meconium concentration; buprenorphine; methadone; pregnant; liquid chromatography-tandem mass spectrometry; opioid-dependant woman
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Methadone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — meconium and urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- exposed mother and child: mother and child who have been exposed to methadone or to buprenorphine during pregnancy
  Interventions: Procedure: Concentrations in Meconium of Buprenorphine and Methadone

INTERVENTIONS:
Procedure: Concentrations in Meconium of Buprenorphine and Methadone — buprenorphine or methadone concentration measurement

SUMMARY:
The aim of this study is to characterize the interest of concentrations in meconium of drugs used for treatment of pregnant opioid-dependent woman as a prognostic factor of time, severity and duration of neonatal abstinence syndrome (NAS). 43 women treated with buprenorphine, 49 with methadone, and their newborns, were included. NAS is assessed by Lipsitz scale. Buprenorphine, norbuprenorphine, methadone, EDDP and morphine are quantified in meconium (one collected immediately after birth, another for 24 to 48 h) by a liquid chromatography-tandem mass spectrometry (LC-MS/MS) method, developed and validated for this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* pregnant women
* Having agreed to participate in the study after information
* Under opioid replacement therapy during pregnancy, in combination or not with other psychotropic drugs or legal or illegal substances.
* Delivery after more than 34 weeks of amenorrhea

Exclusion Criteria:

* Pregnant women not receiving substitution treatment (methadone or buprenorphine).
* Patient under substitution treatment delivering before 34 weeks of amenorrhea
* Patient aged under 18 yrs old
* Patient unable to understand the study (mental deficiency, impairment of consciousness, not French) or not accepting to answer the questionnaires.
* Severe malformation syndrome or chromosomal abnormality in newborn discovered during pregnancy.
* mother's death or newborn's death

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newborns and mothers under opioid replacement therapy during pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
meconium concentration of buprenorphine | variation over time at baseline and 24hrs to 48hrs after birth
meconium concentration of methadone | variation over time at baseline and 24hrs to 48hrs after birth

SECONDARY OUTCOMES:
urine concentration of buprenorphine or methadone | baseline and 24hrs to 48hrs after birth
by the score of Lipsitz, | 4 times a day when the newborn is awake from baseline to 48hrs
  Clinical evaluation of the newborn
screening of other drugs in mother's urine and meconium | baseline and 24hrs to 48hrs after birth

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France